CLINICAL TRIAL: NCT05889117
Title: Neurometabolic Effects of Theta-burst Treatment in Mild Traumatic Brain Injury
Brief Title: Brain Stimulation for Concussion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-110
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Neuropsychological Tests; Traumatic Brain Injury; Post-Concussion Syndrome
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Neuropsychological Tests; Traumatic Brain Injury; Post-Concussion Syndrome; TMS; Theta-burst; Diffusion magnetic resonance spectroscopy
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single group waitlist-control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Waitlist-control-treatment-group (Experimental): After a 2-week control waitlist period, patient receive 30 treatments.
  Interventions: Device: Intermittent theta-burst treatment (iTBS) using MagPro Transcranial Magnetic Stimulator (manufacturer: Magventure)

INTERVENTIONS:
Device: Intermittent theta-burst treatment (iTBS) using MagPro Transcranial Magnetic Stimulator (manufacturer: Magventure) — 3-10 minute sessions of brain stimulation applied to the left dorsolateral prefrontal cortex, up to 10 sessions a day, 30 sessions in total, planned within 2 weeks.
  Other Names: transcranial magnetic stimulation (TMS)

SUMMARY:
The goal of this clinical trial is to test a new type of magnetic brain stimulation in patients with persistent post-concussive symptoms. Participants will undergo detailed MRI scans before and after 30 treatment sessions (of 3-10 minutes each). The main questions the study aims to answer are:

* Will this new type of treatment result in fewer symptoms and better daily functioning?
* What are the effects of this treatment on brain functioning?

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) seems a promising treatment option for patients with persistent post-concussive symptoms (PPCS). Traditional rTMS sessions are relatively long in duration and can be exhaustive for patients with PPCS. Intermittent theta-burst stimulation (iTBS) is a newer and more rapid form of rTMS, which only takes up to 10 minutes per session. However, little is known about the effects of iTBS in patients with PPCS. Furthermore, there is a pressing need for methods that reliably measure the effects of TMS treatments in-vivo. Using diffusion magnetic resonance spectroscopy (dMRS) changes in neural and glial cell morphology can be quantified, which makes it possible to disentangle neurometabolic changes related to neural injury and neuroinflammation, two key elements in the pathophysiology of mTBI.

In the current study, 15 patients with chronic (>3 months after mTBI) PPCS will undergo a total of 30 iTBS sessions. After a baseline scan, patients will enter a 2-week control waitlist period. Following the waitlist control, a pre-treatment scan is acquired, followed by the stimulation sessions, and final post-treatment scan. The scanning protocol includes T1 and T2 imaging, dMRS, multi-shell diffusion MRI (dMRI), as well as a demanding executive function fMRI task, and resting-state fMRI (rs-fMRI). A comprehensive battery of clinical tests will be administered at all time points, which includes cognitive testing, self-report of symptoms and emotional distress. Long-term outcome is determined three months after start of the study.

Specific study aims are:

Aim 1: To determine the effects of a precision-medicine iTBS guided approach applied to the left dorsolateral prefrontal cortex (DLPFC) on clinical recovery in patients with PPCS relative to waitlist control.

Aim 2: To determine the neurometabolic effects of iTBS in both the left and right DLPFC as measured with dMRS in patients with PPS, and to untangle differential effects on pathophysiological processes (e.g., neural plasticity vs. anti-inflammatory effects).

Aim 3: To determine the relationship of these neurometabolic effects and the integrity of major frontoparietal white matter tracts (as measured with dMRI), as well as activation and functional connectivity of key large-scale cognitive and emotional networks (i.e., executive, default mode, and salience network), measured using task-based and resting-state fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Adult age at inclusion 18-64 years.
* mTBI as defined by an altered mental status at time of injury, and LOC of max 30 min, GCS 13-15 (after 30 min), and PTA max 24 hrs.
* Persistent post-traumatic symptoms in chronic phase (>3 months post-injury).

Exclusion Criteria:

* History of developmental, neurological (e.g., epilepsy) or serious mental health disorders (e.g., schizophrenia, bipolar disorder) prior to TBI onset.
* History of a previous substance use disorder except for alcohol, or a currently active substance use disorder (within last 6 months.)
* Contraindications for MRI (e.g., any implanted ferromagnetic materials, claustrophobia, pregnancy) or iTBS (e.g., history of seizures).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-concussive symptoms | Post-treatment (after completion of all sessions, at ~4 weeks), and at 3 months after start of the study for the individual participant. Data will be reported at the conclusion of the study for all participants.
  Rivermead post concussion symptoms questionnaire (16 items, rated 0-4, higher number indicating more symptoms, max score of 64; decrease of the score means improvement of symptoms)
Neurometabolite diffusion related to neuronal function and inflammation | Post-treatment for the individual participant (~4 weeks). Data will be reported at the conclusion of the study for all participants.
  As measured with diffusion MRS (diffusion of neurometabolites computed as the apparent diffusion coefficient (ADC)).

SECONDARY OUTCOMES:
Cognitive functioning | Post-treatment for the individual participant (~4 weeks). Data will be reported at the conclusion of the study for all participants.
  Neuropsychological test scores (attention measured using Stroop interference test: T scores, 0-100, higher scores indicating better performance; processing speed measured using the Symbol search test, also T-scores). Increase in score means clinical improvement.
Functional outcome | At 3 months after start of the study for the individual participant. Data will be reported at the conclusion of the study for all participants.
  Glasgow Outcome Scale Extended (range 1-8, 1=dead, 8=complete recovery; increase in score means clinical improvement).
Brain network functioning | Post-treatment for the individual participant (~ 4 weeks). Data will be reported at the conclusion of the study for all participants.
  As measured with advanced MRI (e.g., improvement on the multimodal attention task can be reflected by a change in percent signal change in the dorsolateral prefrontal cortices of the executive network, which can be either an increase or decrease).

CONTACTS AND LOCATIONS:
Overall Officials: Harm J van der Horn, MD PhD, Principal Investigator — Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical, structural MRI, functional MRI, diffusion MRI, and diffusion MRS data will de-identified, linked to a global unique identifier (GUID) and uploaded to The Federal Interagency Traumatic Brain Injury Research (FITBIR) system. These data will be collected on 15 patients with mild traumatic brain injury. All data are exported in industry-specific, but standardized, formats to promote future research endeavors based on FAIR (Findable, Accessible, Interoperable, and Reusable) Data Principles.